CLINICAL TRIAL: NCT01458665
Title: Arthroscopic Rotator Cuff Repair With Platelet-Rich Plasma (PRP) in Medium to Large Rotator Cuff Tears: A Randomized Controlled Trial
Brief Title: Arthroscopic Rotator Cuff Repair With Platelet-Rich Plasma (PRP) in Medium to Large Rotator Cuff Tears
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hyunchul Jo, Assistant Professor, SMG-SNU Boramae Medical Center, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BRM-11-01
Record Dates: First submitted 2011-10-21; First posted 2011-10-25 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-06

CONDITIONS: Rotator Cuff Tear
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PRP group (Experimental)
  Interventions: Procedure: Arthroscopic rotator cuff repair with PRP
- Conventional group (Placebo Comparator)
  Interventions: Procedure: Conventional arthroscopic rotator cuff repair

INTERVENTIONS:
Procedure: Conventional arthroscopic rotator cuff repair — * Under general anesthesia, the patient was placed in the lazy lateral decubitus position on the operating table.
  * The surgical area was prepared and draped with Betadine.
  * Small stab incisions were made in the creation of 4-5 portals as needed.
  * A scope was explored via the arthroscopic portal into the GH joint & subacromial space.
  * Repair of full thickness rotator cuff tear was done with suture anchors.
  * The skin was closed with Nylon or medical staples.
  * Sterile dressing was applied on surgical wound.
  Arms: Conventional group
Procedure: Arthroscopic rotator cuff repair with PRP — * Under general anesthesia, the patient was placed in the lazy lateral decubitus position on the operating table.
  * The surgical area was prepared and draped with Betadine.
  * Small stab incisions were made in the creation of 4-5 portals as needed.
  * A scope was explored via the arthroscopic portal into the GH joint & subacromial space.
  * Repair of full thickness rotator cuff tear was done with suture anchors.
  * After tying sutures of the medial row, PRP gels were applied on the repair site.
  * The lateral row was secured using suture anchors.
  * The skin was closed with Nylon or medical staples.
  * Sterile dressing was applied on surgical wound.
  Arms: PRP group

SUMMARY:
* The purpose of this study is to compare the clinical and anatomical outcomes of rotator cuff repair with Platelet-Rich Plasma (PRP) and conventional rotator cuff repair in treatment of medium to large rotator cuff tears.
* PRP application to arthroscopic rotator cuff repair would accelerate recovery after arthroscopic rotator cuff repair in terms of pain relief, functional outcomes, overall satisfaction, and enhance structural integrity of repaired tendon.

ELIGIBILITY:
Inclusion Criteria:

medium to large rotator cuff tear as a determined by clinical examination and MR prior to surgery.

Exclusion Criteria:

* previous history of shoulder surgery
* acute trauma
* chronic dislocation
* pyogenic infection
* rotator cuff arthropathy with glenohumeral osteoarthritis and superior migration of the humeral head
* showed abnormal serological test results
* thrombocytopenia (platelets less than 15000 per microliter)
* had been received anti-platelet medication
* psychiatric problems that precludes informed consent or inability to read or write
* other serious problems that preclude participation of the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2011-10; Primary Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Constant-Murley shoulder score | Postoperative 3months
  The Constant score assesses pain, function, ROM, and strength. Pain is allotted a maximum of 15 points, activities of daily living (function)20 points, ROM 40 points, and strength 25 points. The component scores are summated to achieve a maximum possible total score of 100.

CONTACTS AND LOCATIONS:
Overall Officials: Chris H. Jo, M.D., Ph.D, Principal Investigator — Joint & Spine Center, SMG-SNU Boramae Medical Center, Department of Orthopedic Surgery, Seoul National University College of Medicine
Locations (1):
- Joint & Spine Center, SMG-SNU Boramae Medical Center, Department of Orthopedic Surgery, Seoul National University College of Medicine, Seoul, South Korea